CLINICAL TRIAL: NCT04169516
Title: Different Microcirculation Response to Ischemic Injury of Culprit and Non-culprit
Brief Title: Localization of Microvascular Dysfunction
Status: Completed | Type: Observational
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Kyungil Park, Associate professor, Dong-A University
Other Study IDs: 11-95
Record Dates: First submitted 2019-11-14; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Acute Coronary Syndrome
Keywords: microcirculation
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: index of microcirculatory resistance — Physiological parameters of the culprit artery after PCI were determined with the restoration of Thrombolysis in Myocardial Infarction (TIMI) 3 flow. Aortic pressure (Pa), distal intracoronary pressure (Pd), fractional flow reserve (FFR), coronary flow reserve (CFR) and index of microcirculatory resistance (IMR) were measured using a 0.014 coronary temperature and pressure-sensing guidewire (PressureWireCertus, ST. Jude Medical, MN, USA).
  Other Names: 13N-ammonia positron emission tomography

SUMMARY:
Microvascular dysfunction is an independent predictor of poor prognosis. Such response in the culprit vessel is common even after successful revascularization. This study investigated whether the microvascular dysfunction differed between culprit and non-culprit vessels in patients with acute coronary syndrome (ACS) who underwent percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
The prospective study included 115 patients with ACS. In this study, after successful PCI, culprit and non-culprit intracoronary hemodynamic measurements were performed and repeated at 6-month follow-up. 13N-ammonia positron emission tomography (PET) was performed at 6-month follow-up visit to determine absolute myocardial blood flow (MBF). The resistance values of each vessel were calculated using the coronary pressure data and the MBF values obtained from 13N-ammonia PET data. Such physiological measures were compared between culprit and non-culprit vessels in baseline and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Individuals were eligible for inclusion if they underwent PCI for ACS, if the target lesion was found in the proximal or middle segments of a major epicardial coronary artery, and if the lesion was successfully treated with a coronary stent.

Exclusion Criteria:

* a previous infarction other than in the vessel of interest or a history of coronary artery bypass surgery, cardiogenic shock requiring inotropic support, chronic kidney disease requiring renal replacement therapy, hypertrophic cardiomyopathy, collateral flow to the target vessel greater than angiographic grade 1, or statin or ticagrelor use within 1 year.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline index of microcirculatory resistance at 6 months | baseline and 6-month
  Physiological parameters of the culprit artery after PCI were determined with the restoration of Thrombolysis in Myocardial Infarction (TIMI) 3 flow. Index of microcirculatory resistance (IMR) were measured using a 0.014 coronary temperature and pressure-sensing guidewire (PressureWireCertus, ST. Jude Medical, MN, USA). These parameters were then determined for non-culprit vessels.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jo YS, Moon H, Park K. Different Microcirculation Response Between Culprit and Non-Culprit Vessels in Patients With Acute Coronary Syndrome. J Am Heart Assoc. 2020 May 18;9(10):e015507. doi: 10.1161/JAHA.119.015507. Epub 2020 May 15. PMID 32410526